CLINICAL TRIAL: NCT00385268
Title: A Phase II, Double-Blind, Placebo-controlled, Pilot Trial of Acamprosate for the Treatment of Cocaine Dependence
Brief Title: Pilot Trial of Acamprosate for the Treatment of Cocaine Dependence
Acronym: CAMPRAL
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Kyle Kampman, Principal Investigator, University of Pennsylvania
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 803895; P60DA005186 (NIH); DPMC (Other: NIDA); NCT00295451 (obsolete NCT alias)
Record Dates: First submitted 2006-10-06; First posted 2006-10-09 (Estimated); Results first posted 2013-12-31 (Estimated); Last update posted 2020-07-10 (Actual); Status verified 2018-09

CONDITIONS: Cocaine Dependence
Keywords: cocaine
MeSH Terms: conditions — Cocaine-Related Disorders | interventions — Acamprosate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Active medication Acamprosate (Experimental): 1998mg/day for 8 weeks
  Interventions: Drug: acamprosate
- Placebo (Placebo Comparator): placebo pills for 8 weeks
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: acamprosate — 1998 mg/dau fpr 8 weeks
  Other Names: Campral
  Arms: Active medication Acamprosate
Drug: placebo — placebo pills
  Arms: Placebo

SUMMARY:
Trial to determine the safety, efficacy and tolerability of acamprosate for the treatment of cocaine dependence.

DETAILED DESCRIPTION:
The primary objective of the trial is to evaluate the safety, tolerability and efficacy of acamprosate for the treatment of 60 treatment seeking cocaine dependent outpatients. The study will be an exploratory, double-blind, placebo-controlled 9-week trial, with a 2-cell design (30 subjects per cell) in which either 1998 mg/day of acamprosate (666 mg TID) or placebo will be given. Study medications will be given by medical practitioners, trained to provide NIAAA's COMBINE Medical Management. In addition, patients will receive weekly individual psychosocial treatment sessions utilizing Cognitive Behavioral Therapy (CBT) at the University of Pennsylvania Treatment Research Center (TRC).

Primary Hypotheses:

1. Efficacy: Acamprosate-treated subjects will demonstrate less cocaine use during the medication/placebo treatment phase, compared to placebo-treated subjects. Cocaine use will be measured by self-report from the TLFB confirmed with urine assay for benzoylecgonine (BE)
2. Safety and Tolerability: Acamprosate-treated subjects and placebo-treated subjects will report similar rates of adverse events, assessed by weekly evaluations, physical exams and laboratory testing.

Secondary Hypotheses:

1. Acamprosate-treated subjects, compared to placebo-treated subjects, will report less craving for cocaine, measured by lower scores on the Brief Substance Craving Scale (BSCS) (Somoza et al, 1995) and Multiple Choice Procedure (MCP) (Griffiths et al., 1993) during the medication treatment phase.
2. Acamprosate-treated subjects, compared to placebo-treated subjects, will report fewer withdrawal symptoms, measured by the Cocaine Selective Severity Assessment (Kampman et al., 1998).
3. Acamprosate-treated subjects, compared to placebo-treated subjects, will report fewer mood and anxiety symptoms, measured by the Hamilton Depression Rating Scale (HAM-D) (Hamilton, 1967), Hamilton Anxiety Rating Scale (HAM-A) (Hamilton, 1969), and Clinical Global Impression Scale (CGI).
4. Subjects who are highly acamprosate-adherent (>80% pills taken, verified by combining patient report with blister cards) will have more cocaine non-use days during the medication treatment phase, compared to those who are less acamprosate-adherent (<80% pills taken).

ELIGIBILITY:
Inclusion Criteria

1. Male and females 18 years of age or older.
2. Subject meets DSM-IV criteria for current diagnose of cocaine dependence, determined by The Structured Clinical Interview for DSM-IV (SCID-IV).
3. Subject used cocaine in the past 30 days totaling at least $200 worth of cocaine. Cocaine use will be determined by utilizing the modified Timeline Followback, crosschecked with the ASI, which inquires about dollar amounts spent on drug use.
4. Subject lives a commutable distance from the TRC and agrees to attend all research visits, including follow-up visits.
5. Subject speaks, understands, and prints in English.
6. Written informed consent signed by the subject.

Exclusion Criteria

1. Subjects mandated to treatment based upon a legal decision or as a condition of employment.
2. Subjects with evidence of current substance dependence other than cocaine, alcohol or nicotine dependence, as determined by the SCID-IV.
3. Subjects who meets DSM-IV criteria for current alcohol dependence who require a medical alcohol detoxification.
4. Requires treatment with any psychoactive medications, including any anti-seizure medications (with the exception of Benadryl used sparingly, if necessary, for sleep).
5. Has a lifetime DSM-IV diagnosis of bipolar affective disorder, schizophrenia or any psychotic disorder, or organic mental disorder. Has current DSM-IV diagnosis of any other clinically significant psychiatric disorder that will interfere with study participation, as determined by the study physician or PI (Drs. Kyle Kampman, Charles Dackis and Helen Pettinati).
6. Female subjects who are pregnant or lactating, or female subjects of childbearing potential who are not using acceptable methods of birth control. Acceptable methods of birth control include: barrier (diaphragm or condom) with spermicide, intrauterine progesterone contraceptive system, levonorgestrel implant, medroxyprogesterone acetate contraceptive injection, and oral contraceptives.
7. Clinical laboratory tests (CBC, blood chemistries, urinalysis) outside normal limits that are clinically unacceptable to the Principal Investigator. EKG-1st degree heart block, sinus tachycardia, left axis deviation, and nonspecific ST or T wave changes are allowed; liver function tests [LFTs] < 5 x ULN are acceptable. Eligibility will be determined by most recent lab results collected prior to randomization.
8. Subjects with impaired renal function as indicated by corrected creatinine clearance below 80 ml/min/70 kg as determined by the modified Cockcroft equation (Center for Disease Control, 1986).
9. Subjects who have any disease of the gastrointestinal tract, liver or kidneys that could result in a possibility of altered metabolism or excretion of the study drug. As it is not possible to enumerate the many conditions which might impair absorption, metabolism, or excretion, the investigators will be guided by evidence such as: History of major gastrointestinal tract surgery (gastrectomy, gastrostomy, bowel resection, etc) or a history of an active peptic ulcer or chronic disease of the GI tract (ulcerative colitis, regional enteritis, or gastrointestinal bleeding).
10. History of significant heart disease (an arrhythmia which required medication, angina pectoris, documented history of myocardial infarction, or heart failure).
11. Known hypersensitivity to acamprosate.
12. Subjects having participated in any investigational drug trial within 30 days prior to randomizing into the study.
13. Subjects with any serious illnesses that may require hospitalization during the study, as determined by the study physician or PI (Drs. Kyle Kampman, Charles Dackis and Helen Pettinati).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2006-11; Primary Completion 2008-05 (Actual); Study Completion 2008-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Helen Pettinati, Ph.D., Principal Investigator — University of Pennsylvania
Locations (1):
- University of Pennsylvania, Philadelphia, Pennsylvania, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Acamprosate: 1998mg/day for 8 weeks
  Cognitive Behavioral Therapy : Weekly individual psychosocial treatment sessions.
  acamprosate : 1998 mg/dau fpr 8 weeks
- Placebo: placebo pills for 8 weeks
  Cognitive Behavioral Therapy : Weekly individual psychosocial treatment sessions.
  placebo : placebo pills
Period: Overall Study
Arm/Group | Acamprosate | Placebo
Started | 34 | 26
Completed | 18 | 18
Not Completed | 16 | 8

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Acamprosate | Placebo | Total
Number analyzed (Participants) | 34 | 26 | 60
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 34 | 26 | 60
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 45.3 (8.8) | 46.1 (7.7) | 45.5 (7.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 6 | 15
  Male | 25 | 20 | 45
Region of Enrollment [Number; unit: participants]
  United States | 34 | 26 | 60

OUTCOME MEASURES:

1. Primary Outcome: Cocaine Use Over the Eight Week Trial as Measured by Twice Weekly Urine Drug Screen
Description: cocaine abstinent weeks determined by all negative urine drug screens in each week (2 urine drug screens per week)
Time Frame: 8 weeks
Measure: Mean (Standard Deviation); unit: cocaine abstinent weeks
Arm/Group | Acamprosate | Placebo
Number analyzed (Participants) | 34 | 26
cocaine abstinent weeks | 1.3 (2.3) | 1.2 (2.3)
Statistical Analysis 1: Comparison: Acamprosate vs Placebo; Test type: Superiority; p = 0.44, GEE model of repeated measures; GEE on repeated binary indicators of BE positive / negative test; Odds Ratio (OR) = 1.68, 95% CI 2-sided [0.55 to 5.14]

ADVERSE EVENTS:
Arm/Group | Acamprosate | Placebo
Serious Adverse Events (participants affected / at risk) | 0/34 | 0/26
Other Adverse Events (participants affected / at risk) | 13/34 | 13/26
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Acamprosate (N=34) | Placebo (N=26)
Aches and Pains (General disorders) | 13 | 13

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No